CLINICAL TRIAL: NCT00894907
Title: EAGLE: Early Goal-directed Volume Resuscitation in Severe Acute Pancreatitis: A Randomised Multi-centre Study
Brief Title: Early Goal-directed Volume Resuscitation in Severe Acute Pancreatitis
Acronym: EAGLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DFG: HU 1707/2-1
Record Dates: First submitted 2009-05-06; First posted 2009-05-07 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Acute Pancreatitis
Keywords: Severe pancreatitis; acute pancreatitis; haemodynamic monitoring; PiCCO
MeSH Terms: conditions — Pancreatitis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PiCCO-group (Experimental): Insertion of an arterial PiCCO catheter. Resuscitation using crystalloids and/or colloids according to PiCCO-parameter-guided algorithm
  Interventions: Other: PiCCO-parameter-guided volume resuscitation
- 2 (Other): Control: Haemodynamic management without ITBI and ELWI using any other haemodynamic monitoring tool, with the exception of the PiCCO-system.
  Interventions: Other: Control-group

INTERVENTIONS:
Other: PiCCO-parameter-guided volume resuscitation — Insertion of an arterial PiCCO catheter. Resuscitation using crystalloids and/or colloids with the following goals:
  ITBI: 850-1000 ml/sqm, if ELWI <=12*ml/kg; ITBI 750-850 ml/sqm, if ELWI >12*ml/kg and/or PaO2:FiO2 <200 (*ELWI<=12ml/kg, if MAP>65mmHg without catecholamines; ELWI<=14ml/kg, if catecholamines required for MAP>65mmHg); SVV<10% (only in controlled ventilation and sinus rhythm); MAP>65mmHg (MAP: Mean Arterial Pressure); IAPP >60mmHg (IAPP: Intra-abdominal Perfusion Pressure)
  Arms: PiCCO-group
Other: Control-group — Haemodynamic management without ITBI and ELWI using any other haemodynamic monitoring tool, with the exception of the PiCCO-system.
  Main haemodynamic goals: CVP 8-12 mmHg; MAP >65mmHg;IAPP >60mmHg
  Arms: 2

SUMMARY:
Acute pancreatitis (AP) is a common disorder with rising incidence varying between 35 and 80 per 100,000 in Europe and the USA. About 15% of patients develop necrotizing pancreatitis (NP) with a mortality of up to 42% and frequently prolonged hospitalisation in the survivors. Despite a fulminant pathophysiology comparable to that of sepsis, the management of NP is still re-active, symptomatic and mainly based on paradigms with low grade evidence. In sepsis beneficial effects of early goal-directed fluid resuscitation resulting in reduced mortality have been clearly shown. With regard to these data and several studies of NP demonstrating the deleterious effects of fluid loss and haemoconcentration within the first 24h after admission, early goal-directed fluid resuscitation has the potential of improving outcome also in NP. Therefore, it is the aim of this RCT to demonstrate beneficial effects of early goal-directed resuscitation using an algorithm based on modern haemodynamic parameters such as Intra-thoracic Blood Volume Index (ITBI), Extravascular Lung Water Index (ELWI) and Stroke Volume Variation (SVV) which can be easily and safely obtained due to recent progress in haemodynamic monitoring. The algorithm is aimed at maintaining adequate resuscitation (ITBI, SVV) as well as preventing pulmonary over-hydration (ELWI).The use of a similar algorithm in cardiac surgery patients resulted in a significant reduction in catecholamine use, lactate levels, duration of ventilation and ICU stay.

DETAILED DESCRIPTION:
Resuscitation using crystalloids and/or colloids with the following goals:

ITBI: 850 -1000 ml/sqm, if ELWI <=12*ml/kg 750 - 850 ml/sqm, if ELWI >12*ml/kg and/or PaO2:FiO2 <200

*ELWI <=12ml/kg, if MAP>65mmHg without catecholamines <=14ml/kg, if catecholamines required for MAP>65mmHg SVV <10% (only in controlled ventilation and sinus rhythm) MAP >65mmHg (MAP: Mean Arterial Pressure) IAPP >60mmHg (IAPP: Intra-abdominal Perfusion Pressure)

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of pancreatitis:

   * Typical pain
   * Increase in serum lipase or amylase
2. Onset of abdominal pain within <=48h before admission
3. APACHE II >= 8
4. Evidence of >= 1 predictor of severe pancreatitis:

   * Haematocrit >44% (male) or >40% (female), respectively
   * Blood glucose > 125 mg/dl;
   * CRP >= 10 mg/dl;
   * Age > 55 years;
   * Leukocytes >= 16 G/L
   * GOT > 250 U/L;
   * LDH > 350 U/L
   * Calcium < 2,0 mmol/L
   * CK > upper normal range
   * Balthazar-score(CT classification) Grade C-E
   * Any organ failure

Exclusion Criteria:

1. Pregnancy
2. NYHA >II
3. Pre-existing disease with life expectancy < 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2009-08-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Increase in APACHE II >=4 within 4 days as compared to baseline (admission to ICU) | 4 days after admission to the ICU

SECONDARY OUTCOMES:
Mortality | ICU-, 28-days- and in hospital mortality
APACHE-II-Score | 4d; 7d; 28d
Number of ICU-days | Admission to transfer or death
Percentage of organ failure within each group | Time of ICU-stay

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Medical Department; Klinikum Rechts der Isar, Munich, Germany

REFERENCES:
- [Result] Huber W, Umgelter A, Reindl W, Franzen M, Schmidt C, von Delius S, Geisler F, Eckel F, Fritsch R, Siveke J, Henschel B, Schmid RM. Volume assessment in patients with necrotizing pancreatitis: a comparison of intrathoracic blood volume index, central venous pressure, and hematocrit, and their correlation to cardiac index and extravascular lung water index. Crit Care Med. 2008 Aug;36(8):2348-54. doi: 10.1097/CCM.0b013e3181809928. PMID 18596637